CLINICAL TRIAL: NCT01765699
Title: Predicting Poor Outcomes After Primary Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 3878
Record Dates: First submitted 2012-12-31; First posted 2013-01-10 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary knee arthroplasty: Patients with osteoarthritis of the knee undergoing primary knee arthroplasty
  Interventions: Device: Primary knee arthroplasty

INTERVENTIONS:
Device: Primary knee arthroplasty — Patients undergoing primary knee arthroplasty

SUMMARY:
Aim To identify through data analysis key patients, surgeon and operative dependent variables which will improve the performance of knee replacement for primary osteoarthritis

Research Question

1. Can the investigators identify association between outcomes and patients characteristics using existing (already collected) datasets
2. What are the characteristics of patients with poor outcome after knee replacement
3. What can be done to improve the outcome of patients at risk of poor results

DETAILED DESCRIPTION:
This is a retrospective analysis of a prospectively collected single centre database.

ELIGIBILITY:
Inclusion Criteria:

* Primary knee arthroplasty
* Osteoarthritis

Exclusion Criteria:

* No consent for joint registry data collection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone primary knee arthroplasty in our centre.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in PROMS | 1,2,3 and 5 Years post op

CONTACTS AND LOCATIONS:
Overall Officials: Craig Gerrand, Principal Investigator — Consultant Orthopaedic Surgeon; David Deehan, Study Director — Consultant Orthopaedic Surgeon